CLINICAL TRIAL: NCT02454309
Title: A Randomised, Double-blind, Placebo Controlled Trial Evaluating the Effectiveness of a Cranberry Concentrate (CranrichTM) in Preventing Recurrent Urinary Tract Infections in Adult Women
Brief Title: Cranberry for the Prevention of Urinary Tract Infections
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H15-00892
Record Dates: First submitted 2015-05-22; First posted 2015-05-27 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cranberry concentrate (Experimental): Each capsule contains 500 mg of cranberry powder at a concentration ratio of 36:1 (36 grams of cranberries equals 1 gram of concentrate)
  Interventions: Dietary Supplement: Cranberry concentrate
- Placebo (Placebo Comparator): A capsule containing control formulation
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cranberry concentrate
  Other Names: Cranrich (™)
  Arms: Cranberry concentrate
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
This study aims to determine whether a cranberry concentrate reduces recurrent urinary tract infections (UTIs) in women. Approximately 150 adult women will be recruited to participate in this study. Subjects will be randomized to either the cranberry supplement or placebo treatment for 12 months. Subjects and investigators will be blinded to which supplement they are taking.

DETAILED DESCRIPTION:
Participants will be randomized to receive either a cranberry concentrate or placebo. Participants, study staff and investigators will remain blinded until after the dataset has been cleaned. At the baseline visit participants will be instructed to consume the assigned supplement twice daily for 12 consecutive months. A calendar will be provided to record compliance, recurrent UTIs and any side effects. Participants will be phoned/texted each month to encourage participation. Additional study visits will be completed at 3 months, 6 months and 9 months to collect information on recurrent UTIs and adherence. A urine sample will be collected from participants at each visit to test for pregnancy and the presence of an undetected UTI. Supplements will be distributed at each visit for the following 3-month study period and the last bottle of unused product returned. At the 12-month visit, participants will complete an end-line questionnaire and return their supplement bottle in addition to the calendar and side effect diary. If participants withdraw from the study, they will be encouraged to return at 12 months to complete a survey to allow for intent-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* Females who have had at least 2 clinical-diagnosed symptomatic UTIs in the year preceding
* Can communicate in English

Exclusion Criteria:

* Current UTI
* Pregnant or breastfeeding or planning a pregnancy in the next 12 months
* known allergy or intolerance to cranberry-containing products
* A history of renal stones and/or renal transplantation
* Any immunosuppressive disease or other medical conditions that could potentially interfere with outcomes
* Current use of corticosteroid, anticoagulant, antidepressants or mood stabilizing medications or other medications that may interact with the supplement
* Intermittent or indwelling catheterization
* Any anatomic abnormalities of the urinary tract
* The use of any antibiotics within 2 weeks before study entry
* The use of any natural health products, including herbs, homeopathic products, or other forms of cranberry supplements within 2 weeks before study entry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Number of urinary tract infections | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- The University of British Columbia, Vancouver, British Columbia, Canada